CLINICAL TRIAL: NCT01024153
Title: Active Video Games and Sustainable Physical Activity
Acronym: Exergames
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Thomas Baranowski, Professor of Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CA-140670
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Physical Inactivity in Children
Keywords: active video games; children; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active video game play (Experimental)
  Interventions: Behavioral: Active video game play

INTERVENTIONS:
Behavioral: Active video game play — Children will get a Wii video game console and one game at week one and another at week 7. We will monitor their video game play and physical activity during this time.

SUMMARY:
The purpose of this study is to test the effect of active video game play on physical activity of 9-13 year old children in their natural home environments. We observe how much physical activity children engage in after receiving two different active Wii video games and for how long they play. Active video games offer promise of minimizing children's physical inactivity.

DETAILED DESCRIPTION:
The study aims to investigate (1) the temporal trajectory from point of accession of active and inactive video game play in the home environment, (2) the effect of active video game play on overall physical activity and BMI, (3) effects of motivational variables, perceived neighborhood safety, media parenting practices and the home media environment on game play, and (4) what video game characteristics encourage sustainability of play.

Eighty children and their primary caregivers will be recruited to participate in and randomly assigned to the approximately 12 week study. Participating families will be given a Wii* video game console, Wii accessories necessary to play the games and two active or inactive video games**: one at the beginning of the first 6-week period and one at the beginning of the second 6-week period. PA levels of participating children will be measured using accelerometry the week prior to the introduction of the video game (baseline) and on weeks 1, 6, 7, and 12. They will keep a log of video game play on weeks 1, 6, 7 and 12. Objective video game play time will be transcribed at the end of week 12 from calendar stored in the Wii console. Height, weight, waist circumference, triceps skinfold will be measured prior to beginning study (baseline), and weeks 6 and 12. Questionnaires designed to examine the motivation to play a video game (end of weeks 6 and 12) and brief (about 15 minutes) qualitative interview on the children's experiences with the games (end of weeks 6 and 12) will be administered. Parents will complete baseline, week 6 and week 12 questionnaires about their family and child.

*The Wii console has been chosen for this project as it is the platform for the majority of currently popular active video games and it also automatically stores information on name of game played and duration of game play for each play period in a day based calendar. This provides an objective measurement of game use within the family overall, which cannot be modified by the user and can only be deleted by resetting the system.

**To allow reasonably free choice of videos and close replication of the natural setting, the two video games given to a family will be chosen by the 9-12 year-old participant from a selection of either inactive or active video games (depending on group assignment). The Wii video games selected for this study are all rated E (Everyone) by the Entertainment Software Rating Board (E have content suitable for ages 6 and older) and were chosen based on current popularity and review of market rankings. The selected Wii video games include:

Inactive Wii video games: Madden NFL 10, Mario Kart Wii, Super Mario Galaxy and Super Mario Galaxy 2, Disney Sing It, Band Hero, Mario Party 8, Animal Crossing: City Folk, NBA 2K10, New Super Mario Brothers, Sim Animals Africa, Super Paper Mario and Endless Ocean 2: Beautiful Ocean.

Active Wii video games: Wii Sport Resort, Wii Sport, Wii Fit, Wii Play, EA Sports Active, Mario and Sonic at the Olympic Games, Dance, Dance Revolution, Active Life: Extreme Challenge, Academy of Champions, Summer Sports 2: Island Sports Party, and Super Monkey Ball Step and Roll.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 9-12 years old.
* Child and family are able to speak, understand, read and write English.
* No medical problems, including epileptic seizures, that would prevent child from playing inactive or active video games.
* No family history of epileptic seizures.
* Parents will allow child to play our video games.
* Household does not currently has a Wii video game console.
* Baseline visit activity monitor wear will be a compliance criterion for moving forward in the study. Although we ask for 7 days of data, if they return 5 complete days, then they meet the criteria. Without 5 complete days, they are dropped before randomization and thus before receiving the Wii. If we cannot get 5 or 7 days at baseline, it is unlikely that we will get 5 of 7 days at ensuing assessments (based on our 10+ years experience of collecting this type of data).

Exclusion Criteria:

* Children not between the ages of 9-12 years old.
* Child having epilepsy (since playing video games may lead to seizures among those with epilepsy).
* Family history of epileptic seizures.
* Household members not able to speak, understand, read and write English.
* Other medical problems that prevent child from playing inactive or active video games.
* Parents will not allow child to play our video games.
* Household currently has a Wii video game console.
* Child not wearing nor completing the initial baseline 7 day, minimum 800 minutes per day, activity monitor data collection.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
increased physical activity | 4 months

SECONDARY OUTCOMES:
BMI | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Nutrition Research Center, Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] O'Connor TM, Chen TA, Baranowski J, Thompson D, Baranowski T. Physical activity and screen-media-related parenting practices have different associations with children's objectively measured physical activity. Child Obes. 2013 Oct;9(5):446-53. doi: 10.1089/chi.2012.0131. Epub 2013 Sep 12. PMID 24028564
- [Derived] Baranowski T, Abdelsamad D, Baranowski J, O'Connor TM, Thompson D, Barnett A, Cerin E, Chen TA. Impact of an active video game on healthy children's physical activity. Pediatrics. 2012 Mar;129(3):e636-42. doi: 10.1542/peds.2011-2050. Epub 2012 Feb 27. PMID 22371457